CLINICAL TRIAL: NCT06385314
Title: The Effect of Removal of Fixed Partial Dentures on the Grade of Dental Anxiety and State Anxiety a Cross Sectional Study
Brief Title: A Cross Sectional Study on Dental Anxiety and State Anxiety Related to Removal of Fixed Partial Dentures
Status: Completed | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Sponsor
Other Study IDs: Degirmenci1499
Record Dates: First submitted 2024-04-04; First posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Dental Anxiety
MeSH Terms: interventions — Quality of Life

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Oral examination: remove of fixed partial denture for oral examination
  Interventions: Other: Collecting data with oral health related quality of life, dental anxiety and state anxiety
- Denture renewal: remove of fixed partial denture for denture renewal
  Interventions: Other: Collecting data with oral health related quality of life, dental anxiety and state anxiety
- Root canal treatment: remove of fixed partial denture for root canal treatment
  Interventions: Other: Collecting data with oral health related quality of life, dental anxiety and state anxiety
- Tooth extraction: remove of fixed partial denture for tooth extraction
  Interventions: Other: Collecting data with oral health related quality of life, dental anxiety and state anxiety
- Periodontal treatment: remove of fixed partial denture for periodontal treatment
  Interventions: Other: Collecting data with oral health related quality of life, dental anxiety and state anxiety
- Composite filling restoration: remove of fixed partial denture for composite filling restoration
  Interventions: Other: Collecting data with oral health related quality of life, dental anxiety and state anxiety

INTERVENTIONS:
Other: Collecting data with oral health related quality of life, dental anxiety and state anxiety — Collecting data through surveys regarding the patient's oral health related quality of life, dental anxiety and state anxiety before the fixed partial dentures that need to be removed for various clinical reasons are removed.

SUMMARY:
This study aims to evaluate the effect of the clinical removal of fixed partial dentures (FPDs) on oral health-related quality of life (OHRQoL) and the anxiety values of individuals and to determine the risk factors of high anxiety levels. 300 participants were included in this study. Six different reasons for the clinical removal of FPDs (oral examination, denture renewal, root canal treatment, tooth extraction, periodontal treatment, and composite filling restoration) were defined. Questions pertaining to the United Kingdom Oral Health-Related Quality-of-Life Measure (OHQoL-UK), the Modified Dental Anxiety Scale (MDAS), and the Spielberger State-Trait Anxiety Inventory - State (STAI-S) and Trait (STAI-T) were answered.

DETAILED DESCRIPTION:
Data were obtained by questionnaires (United Kingdom Oral Health-Related Quality-of-Life Measure, the Modified Dental Anxiety Scale, the Spielberger State-Trait Anxiety Inventory - State and Trait) after written consent was obtained from all participants. The United Kingdom Oral Health-Related Quality-of-Life Measure (OHQoL-UK) scale is a Likert-type scale, which evaluates the effects of individuals' OHRQoL on 16 main areas in four different categories (symptoms, physical condition, psychological status, and social status) in both positive areas and negative areas, where "1" indicates a very bad impact, "2" denotes a bad effect, "3" represents no effect, "4" indicates a good effect and "5" denotes a very good impact. The minimum and maximum scores can be recorded: 2-10 for the symptom category, 5-25 for the physical condition category, 5-25 for the psychological state category, and 4-20 for the social status category, while the total OHQoL-UK score can be recorded as 16-80. A high OHRQoL score indicates a high quality of life in the relevant category. The Modified Dental Anxiety Scale (MDAS) measures dental anxiety with five questions. The total score can be obtained by adding the scores obtained from five different answer options ranging from 1 (not anxious) to 5 (extremely anxious) in response to the answers given to the five questions about dental anxiety. The total scores of MDAS, which ranged from 5-25, can be divided into two categories "no dental anxiety to moderate dental anxiety" (5-18) and "high dental anxiety" (19-25) points. Spielberger State-Trait Anxiety Inventory has two subscales state anxiety- STAI-S and trait anxiety STAI-T. STAI- state anxiety, measures subjective feelings of apprehension, 'anxious' expectation. STAI- trait anxiety, measures individual differences in anxiety proneness. The STAI consists of 40 items, 20 for each subscale. Items are ordered on a Likert scale from 1 (not at all/almost never) to 4 (very much so/almost always), and some items are reverse-scored. Individuals are asked to indicate how they feel "right now, at this moment" for the STAI-state and how they "generally feel" for the STAI-trait. State (STAI-S) and Trait (STAI-T) scores are obtained by the reverse expressions subtracted from the score of the direct expressions and adding the constant 50 to the state score and the constant 35 to the trait score. A high STAI-S and STAI-T scores indicate a high level of anxiety. Individuals with scores ≥45 on the STAI-S and STAI-T scales can be classified as having high anxiety.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals between the ages of 30 and 65, individuals who are literate and have documented evaluations,
2. Individuals who do not have any physical and psychological health problems,
3. Individuals who do not receive any psychiatric treatment and do not use anxiolytic drugs
4. Individuals who have metal framework porcelain FPDs that need to be removed and are coming in for their removal appointments Individuals who do not have temporomandibular joint problems and neuromuscular disease

Exclusion Criteria:

1. Individuals who have a psychological or psychiatric disorder and use medication,
2. Individuals who have implant-supported FPDs,
3. Individuals who have all-ceramic FPDs or removable dentures,
4. Individuals who have pain that requires emergency intervention
5. Individuals who do not want to be a participant

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population of this cross-sectional study was formed from volunteer participants who presented to the clinic of the Faculty of Dentistry of University between September 2022 and December 2023 and had fixed partial dentures that needed to be removed.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2022-09-05 (Actual); Primary Completion 2023-11-25 (Actual); Study Completion 2023-12-29 (Actual)

PRIMARY OUTCOMES:
United Kingdom Oral Health-Related Quality-of-Life Measure | baseline
  United Kingdom Oral Health-Related Quality-of-Life scale evaluates the effects of individuals' oral health related quality of life.
  Minimum total United Kingdom Oral Health-Related Quality-of-Life scale can be 16. Maximum total United Kingdom Oral Health-Related Quality-of-Life scale score can be 80. Higher scores means a better outcome.
Modified Dental Anxiety Scale | baseline
  Modified Dental Anxiety Scale evaluates dental anxiety of individuals. Minimum total Modified Dental Anxiety Scale score can be 5. Maximum total Modified Dental Anxiety Scale score can be 25. Higher scores means a worse outcome.
Spielberger State Anxiety Inventory | baseline
  Spielberger State Anxiety Inventory evaluates state anxiety of individuals. Minimum total Spielberger State Anxiety Inventory score can be 20. Maximum total Spielberger State Anxiety Inventory score can be 80. Higher scores means a worse outcome. The scores ≥45 on the Spielberger State Anxiety Inventory is classified as having high state anxiety.
Spielberger Trait Anxiety Inventory | baseline
  Spielberger Trait Anxiety Inventory evaluates trait anxiety of individuals. Minimum total Spielberger Trait Anxiety Inventory score can be 20. Maximum total Spielberger Trait Anxiety Inventory score can be 80. Higher scores means a worse outcome. The scores ≥45 on the Spielberger Trait Anxiety Inventory is classified as having high trait anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Kubra Degirmenci, Dr, Principal Investigator — Kubra Degirmenci Faculty of Dentistry Department of Prosthodontics
Locations (1):
- Kubra Degirmenci, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No